CLINICAL TRIAL: NCT04093648
Title: T Cells co- Expressing a Second Generation Glypican 3-specific Chimeric Antigen Receptor With Cytokines Interleukin-21 and 15 as Immunotherapy for Patients With Liver Cancer
Brief Title: T Cells co- Expressing a Second Generation Glypican 3-specific Chimeric Antigen Receptor With Cytokines Interleukin-21 and 15 as Immunotherapy for Patients With Liver Cancer (TEGAR)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The key elements of this study were incorporated into another study.
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Andras Heczey, Assistant Professor, Baylor College of Medicine
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-43874 TEGAR
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma; Hepatoblastoma
Keywords: Hepatocellular Carcinoma; Hepatoblastoma; GPC3-CAR T cells
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatoblastoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TEGAR T cells + Fludarabine and Cytoxan (Experimental): GPC3-CAR (TEGAR T cells) along with lymphodepleting chemotherapy (Cytoxan and Fludarabine) will be administered to patients with hepatocellular carcinoma.
  Interventions: Genetic: TEGAR T cells; Drug: Cytoxan; Drug: Fludarabine

INTERVENTIONS:
Genetic: TEGAR T cells — Five different dosing schedules will be evaluated. Three to six patients will be evaluated on each dosing schedule. The following dose levels will be evaluated:DL1: 1x10^7/m2 DL2: 3x10^7/m2 DL3: 1x10^8/m2 DL4: 3x10^8/m2 DL5: 1x10^9/m2 If DLTs are observed on DL1, patients will be enrolled on DL0 at 3x10^6/m2 dose.
  The first patient on each dose level has to be 28 days post-CAR T cell infusion before the second patient can be enrolled. The doses are calculated according to the actual number of GPC3-CAR transduced T cells.
  Other Names: GPC3-CAR T cells
Drug: Cytoxan — Cyclophosphamide will be given at a dose of 500 mg/m2/day for 3 days given intravenously
  Other Names: Cyclophosphamide
Drug: Fludarabine — Fludarabine will be given at a dose of 30 mg/m2/day for 3 days given intravenously

SUMMARY:
This study is for patients that have a type of cancer that arises from the liver, either called hepatocellular carcinoma or hepatoblastoma. The cancer has come back, has not gone away after standard treatment or the patient cannot receive standard treatment. This research study will use special immune system cells called TEGAR T cells, a new experimental treatment.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise but have not been strong enough to cure most patients. The investigator found from preclinical research that they can put a new gene into T cells that will help them recognize cancer cells and kill them. In our preclinical studies, several genes were made called a chimeric antigen receptor (CAR), from an antibody called GC33 that recognizes glypican-3, a protein found on almost all hepatocellular carcinoma cells and hepatoblastoma cells (GPC3-CAR). In the laboratory the investigators have been doing research into GPC3-CAR cells. They have selected the GPC3-CAR with the strongest ability to recognize hepatocellular carcinoma or hepatoblastoma cells for this study. This is a safety study where the investigator will be testing the ability of GPC3-CAR cells to identify and kill tumor cells in patients. The investigators also tested the effects of adding the molecule interleukin-15 (IL-15) alone or with another molecule called interleukin-21. The investigators found that IL-15 alone or together with IL-21 can help GPC3-CAR T cells last longer which helps them to kill more tumor cells. In this study the investigator will be testing the ability of GPC3-CAR cells to identify and kill tumor cells in patients. This is a study looking at safety and the investigators will therefore be starting with GPC3-CAR T cells alone in a set of patients. The first set of patients will receive GPC3-CAR T cells that also express IL-15. In the second group, the investigators will evaluate GPC3-CAR T cells that express both IL-15 and IL-21. If the investigators are able to safely give GPC3- CAR T cells, they will increase the dose of the combination cells in other patients. The product or dose level of cells that the participant will receive is based on when they are enrolled on the study.

The GPC3-CAR T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of GPC3-CAR T cells that is safe, to see how long they last in the body, to learn what the side effects are and to see if the GPC3-CAR T cells will help people with GPC3-positive hepatocellular carcinoma or hepatoblastoma.

DETAILED DESCRIPTION:
A maximum of 42 subjects will participate in the treatment part of this study.

The investigators will collect up to 180 mL of the participants blood. The investigators will use this blood to grow T cells. They will grow the T cells and use a retrovirus (a special virus that can carry the GPC3 CAR gene into the T cells) to genetically engineer them. After the CAR gene are put into the T cells, the investigators will make sure that they are able to kill hepatocellular carcinoma or hepatoblastoma cells in the laboratory.

LYMPHODEPLETION CHEMOTHERAPY:

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, participants will receive treatment with cyclophosphamide (Cytoxan) and fludarabine for 3 days before receiving the T-cell infusion. These drugs will decrease the numbers of the participants' T cells before the investigator infuse the GPC3-CAR T cells.

WHAT THE INFUSION WILL BE LIKE:

After making these cells, they were frozen. If the patient agrees to participate in this study, they will be scheduled to be treated, the cells will then be thawed and injected into the participant over 5 to 10 minutes. The participant will receive the GPC3-CAR T CELLS 48-72 hours after completing the chemotherapy. The participant may be pretreated with Tylenol (acetaminophen) and Benadryl (diphenhydramine). Tylenol and Benadryl are given to prevent a possible allergic reaction to the T cell administration.

This is a dose escalation study, which means that investigator does not know the highest dose of GPC3-CAR T cells that is safe. To find out, the investigator will give the cells to at least 3 participants at one dose level. If that is safe, the investigator will raise the dose given to the next group of participants. The dose each patient gets will depend on how many participants get the agent before that patient and how they react. The investigator will tell each patient this information. This will help the patient think about possible harms and benefits. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the Treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

Medical tests before treatment:

* Physical exam and History
* EKG (electrocardiogram) to assess heart function
* Blood tests to measure blood cells, kidney and liver function and blood clotting (INR).
* If the patient is infected with the hepatitis B virus (HBV) they will do a test to measure the levels of the virus
* Pregnancy test (if the patient is a female who can get pregnant)
* Measurements of the patient's tumor by scans (CT/MRI) and the tumor marker alfa-fetoprotein (AFP), if the patient's tumor produces this protein.

Medical tests during and after treatment:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function and blood clotting (INR)
* If the patient is infected with the hepatitis B virus (HBV), the investigator will do a test to measure the levels of the virus
* Measurements of the tumor maker alfa-fetoprotein (AFP), if the patient's tumor produces this protein
* Measurements of the patient's tumor by CT/MRI scans (6 -8 weeks after the infusion)
* Tumor biopsy

FOLLOW-UP STUDIES

The investigators will follow the participant during and after the injections. To learn more about the way the T cells are working in the patient's body, up to 60 mL (12 teaspoons) of blood will be taken from the participant before the chemotherapy, before the T-cell infusion, 3 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional) at 1 week, 2 weeks, 4 weeks, 6 weeks and 8 weeks after the injection, every 3 months for 1 year, every 6 months for 4 years and then every year for the next 10 years. Total time participation for this study will be 15 years.

During the time points listed above, if the T cells are found in the patient's blood at a certain amount an extra 5 mL of blood may need to be collected for additional testing.

The investigator will use this blood to look for the frequency and activity of the cells that they have given ; that is, to learn more about the way the T cells are working and how long they last in the body. The investigator will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because patient's have received cells that have had a new gene put in them, they will need to have long term follow up for 15 years so the investigator can see if there are any long term side effects of the gene transfer.

Once a year, the patient will be asked to have their blood drawn and answer questions about their general health and medical condition. The investigators may ask the patient to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present when the patient enrolled in the study and may request that physical exams and/or laboratory tests be performed if necessary.

In the event that a tumor biopsy is performed for clinical reasons the investigators will request permission to obtain excess sample to learn more about the effects of the treatment on the patient's disease. In the event of death, the investigators will request permission to perform an autopsy to learn more about the effects of the treatment on the patient's disease and if there were any side effects from the cells with the new gene .

In addition, the investigators will obtain tumor biopsy for research purposes only. Associated risk with the biopsy will be discussed with the participant in detail in a procedure specific consent form. The investigators will test the sample to see if the GPC3-CAR T cells can be found in the tumor and what effect they had on the tumor cells.

If the patient develops a second abnormal cancer growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested (if a sample can be obtained).

ELIGIBILITY:
Procurement Eligibility

Inclusion Criteria:

* Histology-proven hepatocellular carcinoma (HCC) which is unresectable, recurrent and/or metastatic OR recurrent or resistant hepatoblastoma (HB)
* Barcelona Clinic Liver Cancer Stage A, B or C
* GPC3-positive HCC or HB
* Age ≥ 1 years
* Karnofsky score >60% (See appendix I)
* Life expectancy >12 weeks
* Child-Pugh-Turcotte score <7 (for patients with cirrhosis only)
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

* Heart failure of Class II-IV and / or B-D per NYHA Criteria
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* History of liver transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Severe previous toxicity from cyclophosphamide or fludarabine

Treatment Eligibility

Inclusion Criteria:

* Histology-proven HCC which is unresectable, recurrent and/or metastatic or relapsed / refractory HB
* Barcelona Clinic Liver Cancer Stage A, B or C
* GPC3-positive HCC or HB
* Age ≥ 1 years
* Life expectancy of ≥ 12 weeks
* Karnofsky score ≥ 60%
* Child-Pugh-Turcotte score < 8
* Adequate organ function:
* clearance (as estimated by Cockcroft Gault) ≥ 60 ml/min
* serum AST< 5 times ULN
* total bilirubin < 3 times ULN for age
* INR ≤1.7
* absolute neutrophil count > 500/microliter
* platelet count > 20,000/microliter (can be transfused)
* Hgb ≥9.0 g/dl (can be transfused)
* Pulse oximetry >90% on room air
* Recovered from acute toxic effects of all prior chemotherapy before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Available autologous transduced CAR T cells
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

* Pregnancy or lactation (for women at child-bearing age, birth control is required)
* Receiving investigational drugs within 2 weeks prior to treatment
* Hepatic encephalopathy
* Uncontrolled infection
* Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* History of liver transplantation
* Heart failure of Class II-IV and / or B-D per NYHA Criteria
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* Severe previous toxicity from cyclophosphamide or fludarabine

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) Rate | Start of lymphodepleting chemotherapy to 4 weeks post T cell infusion
  1. DLT rate will be calculated as the number of patients experiencing a DLT divided by the total number of patients receiving treatment.
  2. The NCI Common Toxicity Criteria V5.X will be used in grading toxicity with the exception of CRS and neurological toxicities that are related to T-cell infusions. CRS and neurological toxicities will be graded according to Appendix VI in the protocol.

SECONDARY OUTCOMES:
Response Rate according | 8 weeks post T-cell infusion
  Response rate will be estimated as the percent of patients whose best response is either complete remission or partial remission using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee and by the Immune-related Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Andras Heczey, MD, Principal Investigator — Baylor College of Medicine